CLINICAL TRIAL: NCT00409955
Title: Randomized Clinical Trial for Lamellar Transplants Using Lyophilized and Optisol Corneas
Brief Title: Lamellar Transplant With Lyophilized Corneas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: University of Sao Paulo (Other); Sorocaba Eye Bank (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP 1536/05
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2006-12-12 (Estimated); Status verified 2006-12

CONDITIONS: Keratoconus
Keywords: Lamellar transplant; Lyophilization; Corneas storage; Keratoconus patients; Best corrected visual acuity < 20/60; Signed the consent inform
MeSH Terms: conditions — Keratoconus

INTERVENTIONS:
Procedure: Lamellar transplant with lyophilized corneas

SUMMARY:
- The goals of this study are to develop a lyophilization method for anterior lamellar transplants in Brasil and to make a comparative analysis among patients transplanted with lyophilized and optisol corneas

DETAILED DESCRIPTION:
* After the development of a techinique to lyophilize corneas, we randomly assingned 20 patients with keratoconus and visual acuity of < 20/60, who signed the consent term and divided them into 2 groups. One group was transplanted with lyophilized corneas and the other group with optisol corneas.
* Patients are being followed for 6 months with visual acuity, refraction, topography, orbscan, pachmetry, ultrasound biomicroscopy and confocal microscopy.
* Results are going to be statistically analysed by SPSS program.

ELIGIBILITY:
Inclusion Criteria:

* Keratoconus patient
* BCVA < 20/60
* No systemic diseases
* Who signed the inform consent

Exclusion Criteria:

* BCVA > 20/60
* Presence of deep opacities
* Systemic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-12; Study Completion 2006-12

PRIMARY OUTCOMES:
Topography
Orbscan
Pachmetry
Ultrasound Biomicroscopy
Confocal Microscopy
Masked Examiner to evaluate transparency and quality of the transplant

CONTACTS AND LOCATIONS:
Overall Officials: Roberta JM Farias, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil